CLINICAL TRIAL: NCT00750269
Title: Seamless Phase I/II Study of Stereotactic Lung Radiotherapy (SBRT) for Early Stage, Centrally Located, Non-Small Cell Lung Cancer (NSCLC) in Medically Inoperable Patients
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Stage I Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0813; CDR0000613524; NCI-2009-01095 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); NCT01317056 (obsolete NCT alias)
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Level 1: 8.0 Gy/FX (Experimental): SBRT 40.0 Gy
  Interventions: Radiation: SBRT 40.0 Gy
- Level 2: 8.5 Gy/FX (Experimental): SBRT 42.5 Gy
  Interventions: Radiation: SBRT 42.5 Gy
- Level 3: 9.0 Gy/FX (Experimental): SBRT 45.0 Gy
  Interventions: Radiation: SBRT 45.0 Gy
- Level 4: 9.5 Gy/FX (Experimental): SBRT 47.5 Gy
  Interventions: Radiation: SBRT 47.5 Gy
- Level 5: 10.0 Gy/FX (Experimental): SBRT 50.0 Gy
  Interventions: Radiation: SBRT 50.0 Gy
- Level 6: 10.5 Gy/FX (Experimental): SBRT 52.5 Gy
  Interventions: Radiation: SBRT 52.5 Gy
- Level 7: 11.0 Gy/FX (Experimental): SBRT 55.0 Gy
  Interventions: Radiation: SBRT 55.0 Gy
- Level 8: 11.5 Gy/FX (Experimental): SBRT 57.5 Gy
  Interventions: Radiation: SBRT 57.5 Gy
- Level 9: 12.0 Gy/FX (Experimental): SBRT 60.0 Gy
  Interventions: Radiation: SBRT 60.0 Gy

INTERVENTIONS:
Radiation: SBRT 40.0 Gy — SBRT delivered in 5 fractions of 8.0 Gy/fraction over 1.5 to 2 weeks for a total of 40.0 Gy
  Other Names: Stereotactic body radiation therapy (SBRT); Stereotactic ablative radiotherapy (SABR)
  Arms: Level 1: 8.0 Gy/FX
Radiation: SBRT 42.5 Gy — SBRT delivered in 5 fractions of 8.5 Gy/fraction over 1.5 to 2 weeks for a total of 42.5 Gy
  Other Names: Stereotactic body radiation therapy (SBRT); Stereotactic ablative radiotherapy (SABR)
  Arms: Level 2: 8.5 Gy/FX
Radiation: SBRT 45.0 Gy — SBRT delivered in 5 fractions of 9.0 Gy/fraction over 1.5 to 2 weeks for a total of 45.0 Gy
  Other Names: Stereotactic body radiation therapy (SBRT); Stereotactic ablative radiotherapy (SABR)
  Arms: Level 3: 9.0 Gy/FX
Radiation: SBRT 47.5 Gy — SBRT delivered in 5 fractions of 9.5 Gy/fraction over 1.5 to 2 weeks for a total of 47.5 Gy
  Other Names: Stereotactic body radiation therapy (SBRT); Stereotactic ablative radiotherapy (SABR)
  Arms: Level 4: 9.5 Gy/FX
Radiation: SBRT 50.0 Gy — SBRT delivered in 5 fractions of 10.0 Gy/fraction over 1.5 to 2 weeks for a total of 50.0 Gy
  Other Names: Stereotactic body radiation therapy (SBRT); Stereotactic ablative radiotherapy (SABR)
  Arms: Level 5: 10.0 Gy/FX
Radiation: SBRT 52.5 Gy — SBRT delivered in 5 fractions of 10.5 Gy/fraction over 1.5 to 2 weeks for a total of 52.5 Gy
  Other Names: Stereotactic body radiation therapy (SBRT); Stereotactic ablative radiotherapy (SABR)
  Arms: Level 6: 10.5 Gy/FX
Radiation: SBRT 55.0 Gy — SBRT delivered in 5 fractions of 11.0 Gy/fraction over 1.5 to 2 weeks for a total of 55.0 Gy
  Other Names: Stereotactic body radiation therapy (SBRT); Stereotactic ablative radiotherapy (SABR)
  Arms: Level 7: 11.0 Gy/FX
Radiation: SBRT 57.5 Gy — SBRT delivered in 5 fractions of 11.5 Gy/fraction over 1.5 to 2 weeks for a total of 57.5 Gy
  Other Names: Stereotactic body radiation therapy (SBRT); Stereotactic ablative radiotherapy (SABR)
  Arms: Level 8: 11.5 Gy/FX
Radiation: SBRT 60.0 Gy — SBRT delivered in 5 fractions of 12.0 Gy/fraction over 1.5 to 2 weeks for a total of 60.0 Gy
  Other Names: Stereotactic body radiation therapy (SBRT); Stereotactic ablative radiotherapy (SABR)
  Arms: Level 9: 12.0 Gy/FX

SUMMARY:
RATIONALE: Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase I/II trial is studying the side effects and best dose of stereotactic body radiation therapy and to see how well it works in treating patients with stage I non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose (MTD) of stereotactic body radiotherapy (SBRT) in medically inoperable patients with centrally located stage I non-small cell lung cancer. (Phase I)
* To estimate the local control rate of SBRT at the MTD in these patients. (Phase II)

Secondary

* To estimate the rates of adverse events (other than dose-limiting toxicity) of ≥ grade 3 that is possibly, probably, or definitely related to treatment and that occurs within 1 year after the start of SBRT in these patients.
* To estimate the rates of late adverse events (i.e., occurs > 1 year after the start of SBRT) in these patients.
* To estimate the local control and progression-free and overall survival rates in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients undergo stereotactic body radiotherapy every 2 days over 1½-2 weeks [total of 5 fractions (FX)] in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months for 2 years, then every 6 months for 2 years, then annually.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage T1-2, N0, M0 disease

    * Tumor size ≤ 5 cm
    * Tumor must be within or touching the zone of the proximal bronchial tree, defined as a volume of 2 cm in all directions around the proximal bronchial tree (i.e., carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus right, and left lower lobe bronchi) OR immediately adjacent to the mediastinal or pericardial pleura (PTV touching the pleura)
    * Hilar or mediastinal lymph nodes ≤ 1 cm AND no abnormal hilar or mediastinal uptake on positron emission tomography (PET) scan are considered N0

      * Mediastinal lymph node sampling by any technique is allowed but not required
      * Patients with > 1 cm hilar or mediastinal lymph nodes on CT scan or abnormal PET scan (including suspicious but nondiagnostic uptake) are eligible provided directed tissue biopsies of all abnormally identified areas are negative for cancer
* Tumor deemed technically resectable, in the opinion of an experienced thoracic cancer surgeon, with a reasonable possibility of obtaining a gross total resection with negative margins, defined as a potentially curative resection (PCR)
* Patient deemed "medically inoperable" due to severe underlying physiological medical problems that would prohibit a PCR, including any of the following:

  * Baseline forced expiratory volume at one second (FEV1) < 40% predicted
  * Postoperative FEV1 < 30% predicted
  * Severely reduced diffusion capacity
  * Baseline hypoxemia and/or hypercapnia
  * Exercise oxygen consumption < 50% predicted
  * Severe pulmonary hypertension
  * Diabetes mellitus with severe end-stage organ damage
  * Severe cerebral, cardiac, or peripheral vascular disease
  * Severe chronic heart disease
* Measurable disease as documented by CT scan or whole-body PET scan within the past 8 weeks

  * Patients with lesions that cannot be visualized by CT scan are not eligible
* Pleural effusion allowed provided it is deemed too small to tap under CT guidance and is not evident on chest x-ray

  * Pleural effusion that appears on chest x-ray is allowed only after thoracotomy or other invasive procedure

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 60 days after completion of study therapy
* No other invasive malignancy within the past 2 years except nonmelanomatous skin cancer or carcinoma in situ of the breast, oral cavity, or cervix

  * Prior lung cancer allowed provided the patient has been disease-free for ≥ 2 years

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the region of the study cancer that would result in overlap of radiotherapy fields
* No prior chemotherapy for the study cancer
* No other concurrent local therapy (including standard-fractionated radiotherapy and/or surgery) or systemic therapy (including standard chemotherapy or biologic targeted agents) specifically intended as treatment for study cancer

  * Local or systemic therapy at the time of disease progression allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-02; Primary Completion 2014-09 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bezjak, MD, MSC, FRCPC, Principal Investigator — Princess Margaret Hospital, Canada; Jeffrey Bradley, MD, Study Chair — Mallinckrodt Institute of Radiology at Washington University Medical Center; Laurie E. Gaspar, MD, MBA, Study Chair — University of Colorado, Denver; Robert D. Timmerman, MD, Study Chair — University of Texas; Elizabeth Gore, MD, Study Chair — Medical College of Wisconsin; Feng-Ming Phoenix Konb, MD, PhD, Study Chair — Georgia Regents University Cancer Center
Locations (58):
- United States (57):
  - Arizona Center for Cancer Care - Peoria, Peoria, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Roy and Patricia Disney Family Cancer Center at Providence Saint Joseph Medical Center, Burbank, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Kansas City, Prairie Village, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Norton Suburban Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - McLaren Cancer Institute, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper CyberKnife Center, Mount Laurel, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Bezjak A, Paulus R, Gaspar LE, Timmerman RD, Straube WL, Ryan WF, Garces YI, Pu AT, Singh AK, Videtic GM, McGarry RC, Iyengar P, Pantarotto JR, Urbanic JJ, Sun AY, Daly ME, Grills IS, Sperduto P, Normolle DP, Bradley JD, Choy H. Safety and Efficacy of a Five-Fraction Stereotactic Body Radiotherapy Schedule for Centrally Located Non-Small-Cell Lung Cancer: NRG Oncology/RTOG 0813 Trial. J Clin Oncol. 2019 May 20;37(15):1316-1325. doi: 10.1200/JCO.18.00622. Epub 2019 Apr 3. PMID 30943123
- [Derived] Levy A, Guckenberger M, Hurkmans C, Nestle U, Belderbos J, De Ruysscher D, Faivre-Finn C, Le Pechoux C. SBRT Dose and Survival in Non-Small Cell Lung Cancer: In Regard to Koshy et al. Int J Radiat Oncol Biol Phys. 2015 Jul 15;92(4):945-6. doi: 10.1016/j.ijrobp.2015.03.032. No abstract available. PMID 26104945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was designed to start at dose level 5. Dose levels 1-4 were in place only to be used if the regimen in general proved too toxic and lower dose levels were needed. No patients were accrued to levels 1-4.
Groups:
- Level 5: 10.0 Gy/FX: SBRT 50.0 Gy
  SBRT delivered in 5 fractions of 10.0 Gy/fraction over 1.5 to 2 weeks for a total of 50.0 Gy
- Level 6: 10.5 Gy/FX: SBRT 52.5 Gy
  SBRT delivered in 5 fractions of 10.5 Gy/fraction over 1.5 to 2 weeks for a total of 52.5 Gy
- Level 7: 11.0 Gy/FX: SBRT 55.0 Gy
  SBRT delivered in 5 fractions of 11.0 Gy/fraction over 1.5 to 2 weeks for a total of 55.0 Gy
- Level 8: 11.5 Gy/FX: SBRT 57.5 Gy
  SBRT delivered in 5 fractions of 11.5 Gy/fraction over 1.5 to 2 weeks for a total of 57.5 Gy
- Level 9: 12.0 Gy/FX: SBRT 60.0 Gy
  SBRT delivered in 5 fractions of 12.0 Gy/fraction over 1.5 to 2 weeks for a total of 60.0 Gy
Period: Overall Study
Arm/Group | Level 5: 10.0 Gy/FX | Level 6: 10.5 Gy/FX | Level 7: 11.0 Gy/FX | Level 8: 11.5 Gy/FX | Level 9: 12.0 Gy/FX
Started | 8 | 8 | 18 | 43 | 43
Completed | 8 (Subjects contributing data to the primary analysis are considered to have completed the study) | 7 | 14 | 38 | 33
Not Completed | 0 | 1 | 4 | 5 | 10
Not completed — Protocol Violation | 0 | 1 | 1 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2
Not completed — Patient too large for positioning | 0 | 0 | 1 | 0 | 0
Not completed — Site error | 0 | 0 | 0 | 1 | 0
Not completed — SBRT plan could not be drawn | 0 | 0 | 0 | 0 | 1
Not completed — Fiducials could not be placed | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients receiving protocol treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Level 5: 10.0 Gy/FX | Level 6: 10.5 Gy/FX | Level 7: 11.0 Gy/FX | Level 8: 11.5 Gy/FX | Level 9: 12.0 Gy/FX | Total
Number analyzed (Participants) | 8 | 7 | 14 | 38 | 33 | 100
Age, Continuous [Median (Full Range); unit: years] | 74 [59 to 81] | 75 [53 to 89] | 72 [59 to 81] | 71 [52 to 87] | 72 [55 to 89] | 72 [52 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 6 | 15 | 13 | 43
  Male | 2 | 4 | 8 | 23 | 20 | 57

OUTCOME MEASURES:

1. Primary Outcome: (Phase I) Maximum Tolerated Dose of Stereotactic Body Radiotherapy (SBRT) as Assessed by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0
Description: Maximum tolerated dose (MTD) defined as dose most closely associated with a 20% probability of experiencing a toxicity <= 1 year from start of SBRT from following dose-limiting toxicities: Gr 3-5 Cardiac: Pericardial effusion, Pericarditis, Restrictive cardiomyopathy; Gr 4-5 GI: Dysphagia, Esophagitis, Esophageal fistula/obstruction/perforation/stenosis/ulcer/hemorrhage; Gr 3-5 Nervous System Disorders: Brachial plexopathy, Recurrent laryngeal nerve palsy, Myelitis; Gr 3-5 Respiratory: Atelectasis (gr 4-5 only), Bronchopulmonary/mediastinal/pleural/tracheal hemorrhage, Bronchial/pulmonary/bronchopleural/tracheal fistula, Hypoxia (provided gr 3 is worse than baseline), Bronchial/tracheal obstruction, Pleural effusion, Pneumonitis, Pulmonary fibrosis; Changes in Pulmonary Function Tests per SBRT Pulmonary Toxicity Scale, Gr 3-5: FEV1 decline, FVC decline; Any Gr 5 adverse event attributed to treatment. Dose level was determined by time-to-event continual reassessment method (TITE-CRM).
Time Frame: From start of SBRT to 1 year
Population: All eligible patients who started study treatment
Measure: Number; unit: Gy/FX
Arm/Group | All Participants
Number analyzed (Participants) | 100
Gy/FX | 12.0

2. Primary Outcome: (Phase II) Primary Tumor Control Rate at the Maximum Tolerated Dose (MTD)
Description: Primary tumor control is defined as the absence of primary tumor failure. Primary tumor failure (PTF) refers to the primary treated tumor after protocol therapy and corresponds to meeting following two criteria: 1) Increase in tumor dimension of 20% as defined above for local enlargement (LE); 2) The measurable tumor with criteria meeting LE should be avid on Positron Emission Tomography (PET) imaging with uptake of a similar intensity as the pretreatment staging PET, OR the measurable tumor should be biopsied confirming viable carcinoma. Marginal Failures (MF) and Involved Lobe Failures were also counted as PTF. The cumulative incidence method was used to estimate primary tumor control rate. The 90% confidence interval for local control was calculated using bootstrapping methods. Per the protocol, only the MTD dose level was to be analyzed. However, due to the quantity of patients enrolled on Dose Level 8 as well as safety concerns, Dose Level 8 was analyzed also.
Time Frame: From start of SBRT to 2 years.
Population: All eligible patients who started study treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Level 8: 11.5 Gy/FX | Level 9: 12.0 Gy/FX
Number analyzed (Participants) | 38 | 33
percentage of participants | 89.4 [81.6 to 97.4] | 87.7 [78.3 to 97]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the state of being alive without progression of disease. A failure is the first of the following: local progression, regional progression, distant metastasis, or death. Progression-free survival was assessed at the maximum tolerated dose using the Kaplan-Meier method to estimate the 2-year survival rate. Arms were not compared/tested.
Time Frame: From randomization to date of death, failure (local, regional or distant) or last follow-up. Analysis occurs after all patients have been potentially followed for 24 months, approximately 7.5 years from the start of the study.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Level 5: 10.0 Gy/FX; Level 6: 10.5 Gy/FX: SBRT delivered in 5 fractions of 10.5 Gy/fraction over 1.5 to 2 weeks for a total of 52.5 Gy
- Level 7: 11.0 Gy/FX: SBRT delivered in 5 fractions of 11.0 Gy/fraction over 1.5 to 2 weeks for a total of 55.0 Gy
Arm/Group | Level 5: 10.0 Gy/FX | Level 6: 10.5 Gy/FX | Level 7: 11.0 Gy/FX | Level 8: 11.5 Gy/FX | Level 9: 12.0 Gy/FX
Number analyzed (Participants) | 8 | 7 | 14 | 38 | 33
percentage of participants | 50.0 [15.2 to 77.5] | 57.1 [17.2 to 83.7] | 57.1 [28.4 to 78.0] | 52.2 [35.3 to 66.6] | 54.5 [36.3 to 69.6]

4. Secondary Outcome: Overall Survival
Description: An event for overall survival is death due to any cause. Overall survival was assessed at the maximum tolerated dose using the Kaplan-Meier method to estimate the 2-year survival rate. Arms were not compared/tested.
Time Frame: From randomization to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 24 months, approximately 7.5 years from the start of the study.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Level 5: 10.0 Gy/FX: SBRT delivered in 5 fractions of 10.0 Gy/fraction over 1.5 to 2 weeks for a total of 50.0 Gy
Arm/Group | Level 5: 10.0 Gy/FX | Level 6: 10.5 Gy/FX | Level 7: 11.0 Gy/FX | Level 8: 11.5 Gy/FX | Level 9: 12.0 Gy/FX
Number analyzed (Participants) | 8 | 7 | 14 | 38 | 33
percentage of participants | 75.0 [31.5 to 93.1] | 57.1 [17.2 to 83.7] | 71.4 [40.6 to 88.2] | 70.2 [52.6 to 82.3] | 72.7 [54.1 to 84.8]

5. Secondary Outcome: Local Progression
Description: Local progression is the same as primary tumor failure (PTF) which refers to the primary treated tumor after protocol therapy and corresponds to meeting both of the following two criteria: 1) Increase in tumor dimension of 20% as defined above for local enlargement (LE); 2) The measurable tumor with criteria meeting LE should be avid on Positron Emission Tomography (PET) imaging with uptake of a similar intensity as the pretreatment staging PET, OR the measurable tumor should be biopsied confirming viable carcinoma. For outcome analysis, Marginal Failures (MF) and Involved Lobe Failures will also be counted as PTF. Local progression was assessed using the cumulative incidence method to estimate the 2-year failure rate. Arms were not compared/tested.
Time Frame: From randomization to date of death, regional failure or last follow-up. Analysis occurs after all patients have been potentially followed for 24 months.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Level 5: 10.0 Gy/FX | Level 6: 10.5 Gy/FX | Level 7: 11.0 Gy/FX | Level 8: 11.5 Gy/FX | Level 9: 12.0 Gy/FX
Number analyzed (Participants) | 8 | 7 | 14 | 38 | 33
percentage of participants | 12.5 [0.5 to 44.5] | 0 [NA to NA] — A confidence interval cannot be computed when the rate is zero, i.e. when there are zero events. | 14.3 [2.1 to 37.7] | 10.6 [3.3 to 22.9] | 12.3 [3.8 to 26.1]

6. Secondary Outcome: Nodal Progression
Description: Regional nodal progression is defined as appearance after protocol therapy of measurable tumor within lymph nodes along the natural lymphatic drainage typical for the location of the treated primary disease only with dimension of at least 1.0 cm on imaging studies (preferably CT scans) within the lung, bronchial hilum, or the mediastinum. Regional nodal progression was assessed using the cumulative incidence method to estimate the 2-year failure rate. Arms were not compared/tested.
Time Frame: From randomization to date of death, regional failure or last follow-up. Analysis occurs after all patients have been potentially followed for 24 months, approximately 7.5 years from the start of the study.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Level 5: 10.0 Gy/FX | Level 6: 10.5 Gy/FX | Level 7: 11.0 Gy/FX | Level 8: 11.5 Gy/FX | Level 9: 12.0 Gy/FX
Number analyzed (Participants) | 8 | 7 | 14 | 38 | 33
percentage of patients | 0 [NA to NA] — A confidence interval cannot be computed when the rate is zero, i.e. when there are zero events. | 0 [NA to NA] — A confidence interval cannot be computed when the rate is zero, i.e. when there are zero events. | 7.1 [0.4 to 28.7] | 5.3 [0.9 to 15.7] | 6.1 [1 to 17.9]

7. Secondary Outcome: Distant Metastases
Description: Distant metastases is defined as the appearance after protocol therapy of cancer deposits characteristic of metastatic dissemination from non-small cell lung cancer. Distant metastases progression was assessed using the cumulative incidence method to estimate the 2-year failure rate. Arms were not compared/tested.
Time Frame: From randomization to date of death, distant failure or last follow-up. Analysis occurs after all patients have been potentially followed for 24 months, approximately 7.5 years from the start of the study.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Level 5: 10.0 Gy/FX | Level 6: 10.5 Gy/FX | Level 7: 11.0 Gy/FX | Level 8: 11.5 Gy/FX | Level 9: 12.0 Gy/FX
Number analyzed (Participants) | 8 | 7 | 14 | 38 | 33
percentage of participants | 0 [NA to NA] — A confidence interval cannot be computed when the rate is zero, i.e. when there are zero events. | 14.3 [0.4 to 50.3] | 14.3 [2.1 to 37.6] | 7.9 [2 to 19.3] | 15.2 [5.4 to 29.5]

8. Secondary Outcome: Rate of Toxicity ≥ Grade 3 (Other Than DLT) Within One Year as Assessed by NCI CTCAE v4.0
Description: Rate of patients developing any treatment-related toxicity during the first year following the start of SBRT that is not among the types considered as a dose-limiting toxicity.
Time Frame: From start of SBRT until 1 year.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Level 5: 10.0 Gy/FX | Level 6: 10.5 Gy/FX | Level 7: 11.0 Gy/FX | Level 8: 11.5 Gy/FX | Level 9: 12.0 Gy/FX
Number analyzed (Participants) | 8 | 7 | 14 | 38 | 33
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 12.1 [2.9 to 24.8] | 16.7 [3.4 to 28.2]

9. Secondary Outcome: Rate of Late Toxicity (i.e., Occurs > 1 Year After the Start of SBRT) of ≥ Grade 3 as Assessed by NCI CTCAE v4.0
Description: Percentage of patients who developed any treatment-related toxicity after the first year following the start of SBRT.
Time Frame: From start of treatment to end of follow-up. Analysis occurs after all patients have been potentially followed for 24 months, approximately 7.5 years from the start of the study.
Population: All eligible patients who started study treatment who were observed more than 1 year after start of SBRT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Level 5: 10.0 Gy/FX | Level 6: 10.5 Gy/FX | Level 7: 11.0 Gy/FX | Level 8: 11.5 Gy/FX | Level 9: 12.0 Gy/FX
Number analyzed (Participants) | 8 | 5 | 12 | 32 | 31
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 16.7 [2.1 to 48.4] | 6.3 [0.8 to 20.8] | 16.1 [5.5 to 33.7]

ADVERSE EVENTS:
Description: Patients experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Level 5: 10.0 Gy/FX | Level 6: 10.5 Gy/FX | Level 7: 11.0 Gy/FX | Level 8: 11.5 Gy/FX | Level 9: 12.0 Gy/FX
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/7 | 2/14 | 9/38 | 7/33
Other Adverse Events (participants affected / at risk) | 7/8 | 7/7 | 13/14 | 34/38 | 27/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Level 5: 10.0 Gy/FX (N=8) | Level 6: 10.5 Gy/FX (N=7) | Level 7: 11.0 Gy/FX (N=14) | Level 8: 11.5 Gy/FX (N=38) | Level 9: 12.0 Gy/FX (N=33)
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Esophageal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Death NOS (General disorders) | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Level 5: 10.0 Gy/FX (N=8) | Level 6: 10.5 Gy/FX (N=7) | Level 7: 11.0 Gy/FX (N=14) | Level 8: 11.5 Gy/FX (N=38) | Level 9: 12.0 Gy/FX (N=33)
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Mitral valve disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 2 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Tricuspid valve disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 4 | 5 | 9
Esophageal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Esophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1
Esophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Esophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Death NOS (General disorders) | 0 | 1 | 1 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 4 | 3 | 6 | 12 | 8
Fever (General disorders) | 1 | 0 | 0 | 2 | 0
Pain (General disorders) | 2 | 0 | 0 | 0 | 2
Bronchial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 2 | 1 | 1 | 2 | 1
Forced expiratory volume decreased (Investigations) | 1 | 2 | 3 | 5 | 1
Investigations - Other (Investigations) | 0 | 0 | 1 | 0 | 0
Vital capacity abnormal (Investigations) | 1 | 1 | 0 | 1 | 0
Weight loss (Investigations) | 1 | 0 | 0 | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Brachial plexopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Myelitis (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3 | 13 | 13
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 3
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 11 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 5 | 11 | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 8 | 7
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5 | 7 | 11
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3 | 13 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 2 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 5 | 7
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.